CLINICAL TRIAL: NCT06529965
Title: Evaluating a Digital Intervention for Alleviating Diabetes-specific Emotional Distress in Adults Living With Type 2 Diabetes Mellitus: Randomized Controlled Trial
Brief Title: Evaluating a Digital Intervention for Alleviating Diabetes-specific Emotional Distress in Adults Living With T2DM
Acronym: EASE-T2DM
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Gaia AG (Industry)
Collaborators: University Hospital Schleswig-Holstein (Other); Philipps University Marburg (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: covivio RCT 2024
Record Dates: First submitted 2024-07-26; First posted 2024-07-31 (Actual); Last update posted 2024-11-08 (Actual); Status verified 2024-11

CONDITIONS: Glucose Metabolism Disorders (Including Diabetes Mellitus); Metabolic Disease; Endocrine System Diseases; Diabetes Mellitus, Type 2
Keywords: type 2 diabetes; covivio; diabetes self-management; digital health application
MeSH Terms: conditions — Glucose Metabolism Disorders; Metabolic Diseases; Endocrine System Diseases; Diabetes Mellitus, Type 2

STUDY DESIGN:
Intervention Model Description: randomized controlled trial with two arms: (i) online intervention in addition to treatment-as-usual versus (ii) treatment-as-usual
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention/Treatment (Experimental): Experimental: covivio + TAU
  Participants allocated to the intervention group will receive access to covivio in addition to treatment as usual (TAU).
  covivio is a digital health application designed for individuals with type 2 diabetes mellitus who suffer from elevated levels of diabetes-specific emotional distress, accessible through a web browser. The application focuses on treatment methods derived from cognitive behavioral therapy (CBT). Topics addressed by covivio are disease literacy, physical activity and exercise, nutrition, stress management, sleep management, mood problems, and social resources.
  The program operates through interactive "dialogues", which are accompanied by illustrations, audio recordings, motivational text messages, worksheets, and summaries. Users are also encouraged to regularly complete short questionnaires to monitor their complaints. Once registered, the program remains accessible for 180 days.
  Interventions: Behavioral: covivio
- Control (No Intervention): No Intervention: TAU
  Participants allocated to the control group will receive access to treatment as usual (TAU).

INTERVENTIONS:
Behavioral: covivio — Participants will receive access to the digital health intervention covivio in addition to TAU.
  Arms: Intervention/Treatment

SUMMARY:
This randomized controlled trial (RCT) with 250 patients suffering from type 2 diabetes mellitus (T2DM) aims to investigate the effectiveness of the self-guided digital therapeutic covivio. Inclusion criteria are: male, female or non-binary; age ≥ 18 years; confirmed diagnosis of T2DM; elevated levels of diabetes-specific emotional distress (Problem Areas in Diabetes [PAID]-20 score ≥ 33); consent to participate; sufficient German language skills. Exclusion criteria are: a diagnosis of type 1 diabetes mellitus (T1DM); current use of continuous glucose monitoring (CGM) as part of one's diabetes treatment; changes or planned changes in medication within 4 weeks before the baseline visit or in the subsequent 6 months; a bariatric operation within 4 weeks before the baseline visit or such an operation planned in the subsequent 6 months; changes or planned changes in psychotherapeutic treatment within 4 weeks before the baseline visit or in the subsequent 6 months. In addition, participants will be excluded from the study if they did not wear the CGM sensor for at least 6 of 7 days at baseline (before randomization), providing a minimum of 96 hours of glucose values including at least 24 hours overnight.

Patients will be randomized and allocated in a 1:1 ratio to either an intervention group, in which they will receive access to covivio in addition to treatment as usual (TAU, n = 125), or to a control group, in which they will receive only TAU (n = 125).

Co-primary endpoints of this trial will be the between-groups difference in the PAID-20 total score in the intervention and control group at six months, adjusted for the PAID-20 baseline score as well as the glucose management indicator (estimated HbA1c) assessed using continuous glucose monitoring devices (for a period of 7 days) at six months, adjusted for the baseline score.

Secondary endpoints will be diabetes self-management skills, body mass index (BMI), and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* male, female or non-binary
* age ≥ 18 years
* diagnosis of T2DM secured via submission of a medical certificate attesting to the presence of at least one of the following ICD-10-GM diagnoses of T2DM: E11.20, E11.30, E11.40, E11.50, E11.60, E11.72, E11.74, E11.80, E11.90
* elevated levels of diabetes-specific emotional distress: cut-off ≥ 33 on the PAID-20
* access to CGM-compatible smartphone
* consent to participate
* sufficient knowledge of the German language

Exclusion Criteria:

* diagnosis of type 1 diabetes mellitus (T1DM)
* change in medication (type, frequency of use or dosage) within 4 weeks before the baseline visit or planned within the subsequent 6 months
* recent or planned bariatric operation within 4 weeks before the baseline visit or within the subsequent 6 months
* change in psychotherapeutic treatment within 4 weeks before the baseline visit or planned within the subsequent 6 months
* current use of continuous glucose monitoring (CGM) as part of one's diabetes treatment
* experiencing problems with the CGM sensor or insufficient CGM data quality at baseline (T0) (i.e., wearing the CGM sensor on less than 6 of 7 days, providing less than a minimum of 96 hours of glucose values, providing less than 24 hours overnight CGM data)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2024-10-09 (Actual); Primary Completion 2026-04-09 (Estimated); Study Completion 2026-04-09 (Estimated)

PRIMARY OUTCOMES:
Diabetes-specific emotional distress | 6 months
  Assessed with the Problem Areas in Diabetes Questionnaire (PAID-20). Total score ranging from 0-100; higher scores indicate higher diabetes-specific emotional distress (worse outcome).
Glucose management indicator | 6 months
  The glucose management indicator (GMI) is an estimation of HbA1c from CGM. It is calculated as follows: GMI (%) = 3.31 + 0.02392 x [mean glucose in mg/dL].

SECONDARY OUTCOMES:
Diabetes-specific emotional distress | 3 months
  Assessed with the Problem Areas in Diabetes Questionnaire (PAID-20). Total score ranging from 0-100; higher scores indicate higher diabetes-specific emotional distress (worse outcome).
Diet self-management skills | 3 months; 6 months
  Assessed with the Diet Subscale of the Summary of Diabetes Self-Care Activities Measure (SDSCA). The diet subscale contains four items and the score may range from 0-28; higher scores indicate higher diet self-management skills (better outcome).
Exercise self-management skills | 3 months; 6 months
  Assessed with the Exercise Subscale of the Summary of Diabetes Self-Care Activities (SDSCA). The exercise subscale contains two items and the score may range from 0-14; higher scores indicate higher exercise self-management skills (better outcome).
Health-related quality of life | 3 months; 6 months
  Quantified with the Assessment of Quality of Life - 8 Dimensions (AQoL-8D). Total score ranging from 0-100; higher scores indicate a higher quality of life (better outcome).
Body mass index (BMI) | 3 months; 6 months
  The BMI will be computed according to the following formula: kg/m2, where kg is a person's weight in kilograms and m2 is their height in meters squared. If necessary, height will be converted into meters and weight will be converted into kilograms.

OTHER OUTCOMES:
Time in range (TIR) derived from CGM | 6 months
  Defined as time spent in the target range between 70 and 180 mg/dL. TIR will be assessed in hours and minutes for a 7-day period, and also expressed as percent.
Mean sensor glucose derived from CGM | 6 months
  Mean sensor glucose will be calculated over the 7 days of glucose measurements.
Coefficient of variation derived from CGM | 6 months
  The coefficient of variation will be used to quantify glycemic variability.

CONTACTS AND LOCATIONS:
Overall Officials: Kamila Jauch-Chara, Dr. med., Principal Investigator — Zentrum für Integrative Psychiatrie, Universitätsklinikum Schleswig-Holstein
Locations (1):
- GAIA AG, Hamburg, Germany

IPD SHARING:
Plan to Share IPD: No